CLINICAL TRIAL: NCT02424513
Title: A Phase 2 Study of Positron Emission Tomography (PET) With [89]Zr-Df-IAb2M in Patients With High-risk Prostate Cancer
Brief Title: A Study of Positron Emission Tomography (PET) With [89]Zr-Df-IAb2M in Patients With High-risk Prostate Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical trial was postponed as a result of restructured business priorities.
Sponsor: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2014-2M-04.00
Record Dates: First submitted 2015-04-14; First posted 2015-04-23 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2015-05

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 89Zr-Df-IAB2M

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- [89Zr]Df-IAB2M (Experimental): A single intravenous infusion of 2.5 mCi of [89Zr]Df-IAB2M in a mass dose of 10 mg.
  Interventions: Radiation: [89Zr]Df-IAB2M

INTERVENTIONS:
Radiation: [89Zr]Df-IAB2M — A single intravenous infusion of 2.5 mCi of [89Zr]Df-IAB2M in a mass dose of 10 mg.

SUMMARY:
This is a prospective, multicenter, open-label, non-randomized study evaluating the ability of [89]Zr-Df-IAb2M to detect local, regional and metastatic prostate cancer confirmed by pathology.

DETAILED DESCRIPTION:
IAB2M is an approximately 80 kDA molecular weight antibody fragment (a "Minibody") chelated with Desferroxamine and radiolabeled with [89]Zr. [89Zr]-Df-IAB2M targets the extracellular domain of Prostate Membrane Specific Antigen (PSMA) expressed on most primary and metastatic prostate cancer lesions.

This is a phase 2, prospective, multi-center, open-label, non-randomized study evaluating the ability of [89]Zr-Df-IAb2M to detect local, regional and metastatic prostate cancer confirmed by pathology in patients with biopsy-proven prostate cancer thought to be candidates for radical prostatectomy and pelvic lymph node dissection who are at high-risk for pelvic lymph node metastasis. These patients may have identified lymphadenopathy on conventional imaging but are considered eligible if still judged to be candidates for radical prostatectomy and lymph node dissection.

ELIGIBILITY:
Inclusion Criteria:

1. Histological diagnosis of prostate adenocarcinoma.
2. Patients considered candidates for radical prostatectomy and pelvic lymph node dissection. These patients may or may not have identified nodal metastasis on conventional imaging but would still be candidates for radical prostatectomy and pelvic lymph node dissection.
3. Patients, who are at high-risk for pelvic lymph node metastasis as defined by a lymph node involvement risk of greater than or equal to 20% using the Briganti nomogram.
4. Age ≥ 18 years.
5. Ability to understand and willingness to sign IRB approved consent form
6. For men of child-producing potential, the use of effective contraceptive methods during the study.

Exclusion Criteria:

1. Treatment or plans for treatment with radiation therapy, surgery, chemotherapy, or investigational therapy between the time of conventional imaging, [89]Zr-Df-IAB2M PET/CT and the surgical resection or biopsy procedures used for the study evaluation.
2. Unwillingness or inability to comply with procedures required in this protocol.
3. Other cancers that might potentially interfere with the reading and interpretation of [89]Zr-Df-IAB2M PET/CT scans.
4. Patients who are currently receiving any other investigational agent.
5. Patients who have had or are currently receiving androgen deprivation therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-03; Primary Completion 2016-03 (Estimated); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of [89]Zr-Df-IAb2M PET/CT for the detection of extraprostatic sites of prostate cancer as confirmed by biopsy and/or surgically resected tissue. | 6 weeks
Specificity of [89]Zr-Df-IAb2M PET/CT for the detection of extraprostatic sites of prostate cancer as confirmed by biopsy and/or surgically resected tissue. | 6 weeks
Positive Predicted Value of [89]Zr-Df-IAb2M PET/CT for the detection of extraprostatic sites of prostate cancer as confirmed by biopsy and/or surgically resected tissue. | 6 weeks
Negative Predicted Value of [89]Zr-Df-IAb2M PET/CT for the detection of extraprostatic sites of prostate cancer as confirmed by biopsy and/or surgically resected tissue. | 6 weeks
Accuracy of [89]Zr-Df-IAb2M PET/CT for the detection of extraprostatic sites of prostate cancer as confirmed by biopsy and/or surgically resected tissue. | 6 weeks

SECONDARY OUTCOMES:
optimal SUVmax and SUVpeak thresholds on [89]Zr-Df-IAb2M PET/CT for discriminating positive and negative tumor pathology results. | 6 weeks
Optimal SUV ratio thresholds on [89]Zr-Df-IAb2M PET/CT for discriminating positive and negative tumor pathology results, where the ratio is calculated using an appropriate reference tissue. | 6 weeks
Sensitivity and specificity of [89]Zr-Df-IAb2M PET/CT compared to the sensitivity and specificity of conventional imaging for the detection of lesions as confirmed by pathology. | 6 weeks
Location and number of positive lesions on [89]Zr-Df-IAb2M PET/CT in subjects with equivocal or negative conventional imaging scans. | 6 weeks
Sensitivity and specificity of [89]Zr-Df-IAb2M PET/CT to identify patients who are positive or negative for metastatic disease as identified by pathology. | 6 weeks
Sensitivity and specificity of IAB2M [89]Zr-Df-IAb2M PET/CT to identify disease as confirmed by pathology individually in each of the resected areas including: left and right external iliac, obturator and internal iliac nodes. | 6 weeks

OTHER OUTCOMES:
Number of Participants with Adverse Events or Serious Adverse Events attributable to [89]Zr-Df-IAB2M administration according to MedDRA/CTCAE v. 4.03 as a measure of safety and tolerability. | 12 weeks
Number of Participants with clinically significant changes in physical examination findings, vital signs, and blood chemistry from screening to follow-up analysis as a measure of safety and tolerability. | 12weeks
Number of Participants with Anti-drug antibody (ADA) in serum due to [89]Zr-Df-IAB2M injection as a measure of safety and tolerability. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: James Eastham, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Washington University, St Louis, Missouri, United States